CLINICAL TRIAL: NCT01782040
Title: Auriculotherapy in the Cares to the Premenstrual Syndrome: Randomized Clinical Trial
Brief Title: Auriculotherapy in the Cares to the Premenstrual Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Sociedade Hospital Samaritano (Other)
Responsible Party: Principal Investigator, Leonice Fumiko Sato Kurebayashi, Leonice Fumiko Sato Kurebayashi, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 35/2010
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; Physical distress; Behavioral changes
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Control Group didn't receive any treatment and it was evaluated at the same time and the same way of interventions group
- Auriculotherapy group (Experimental): The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to treat several kind of diseases using semi-permanent needles in specific points of the auricular pavilion.It was used 6 points: Kidney, Liver, Stomach, Brain Stem, Ovary and Uterus point with semi-permanent needles one time per week for 8 sessions
  Interventions: Other: Auriculotherapy group

INTERVENTIONS:
Other: Auriculotherapy group — It was used semipermanent needles (1.5mm) to stimulate points, once on a week, during 8 sessions.
  Other Names: Auricular acupuncture
  Arms: Auriculotherapy group

SUMMARY:
Premenstrual syndrome (PMS) is a collection of physical and emotional symptoms related to a woman's menstrual cycle. These symptoms occurring only during the luteal phase of the menstrual cycle that are of sufficient severity to interfere with some aspects of life of these women, reflecting also in interpersonal relationships, workplace and in their productivity. For these reasons, this research was conducted with the nursing staff of the Samaritan Hospital in order to verify the effectiveness of auricular acupuncture to alleviate some of the symptoms of PMS.

DETAILED DESCRIPTION:
The chinese auriculotherapy is a intervention used by Chinese Traditional Medicine in order to balance the body energy and to treat several kind of diseases using semipermanent needles in specific points of the auricular pavilion.

ELIGIBILITY:
Inclusion Criteria:

1. Belong to the nursing staff
2. Present at least one behavioral or physical symptom that is self-perceived as related to the symptoms that precede menstruation (irritability, depression, fatigue, headache, breast tenderness, swelling, anxiety, insomnia, crying spells, changes in appetite)
3. Voluntary participation in the study
4. Availability of time for submission to the sessions

Exclusion Criteria:

1. Medical license or vacation during the period of the research.
2. Pregnancy

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Premenstrual syndrome symptoms | after 3 months
  This randomized clinical trial aimed at evaluating the auriculotherapy efficacy to reduce behavioral or physical symptom that is self-perceived as related to the symptoms that precede menstruation (irritability, depression, fatigue, headache, breast tenderness, swelling, anxiety, insomnia, crying spells, changes in appetite)

CONTACTS AND LOCATIONS:
Overall Officials: Leonice FS Kurebayashi, Ms, Principal Investigator — São Paulo University; Rafael FB Homo, Study Chair — University of Sao Paulo; Ana LL Giaponesi, Principal Investigator — Samaritan Hospital; Maria JP Silva, Phd, Study Director — University of Sao Paulo
Locations (1):
- Samaritan Hospital, São Paulo, São Paulo, Brazil